CLINICAL TRIAL: NCT02855216
Title: Comparative Study of the Effects of Two Sub-occipital Techniques on Healthy Subjects With Limited Mobility According to the Flexion-rotation Test
Brief Title: Effects of Two Sub-occipital Techniques on Limited Mobility According to the Flexion-rotation Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Andoni Carrasco, PT, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI16/0147
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Upper Cervical Spine Rotational Hypomobility
Keywords: Physiotherapy; Range of motion; Inhibition sub-occipital techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual technique of sub-occipital inhibition (Experimental): The technique applied to Manual Group was performed with the patient supine position. Physiotherapist in a sitting position at the head of the subject with forearms resting on the table . Suboccipital region was located , and flexing the metacarpophalangeal joints 90º a pressure was made ventrally , relaxing the rest of the head in the heel of the hand.
  The technique was performed for 5 minutes
  Interventions: Other: Manual technique of sub-occipital inhibition
- Self-treatment by way of Occipivot® (Experimental): The technique applied to the Instrumental Group was performed with the patient supine in the same position as the Manual Group . It was previously instructed the subject how to proceed with the cushion Occipivot® , indicating the installation location and method of affixing , correcting him if the application was inadequate. The subject placed the cushion Occipivot® under the suboccipital region and told him he had to stay in that position for 5 minutes. A physiotherapist warned the patient at the end of the application time so that the subject had to be aware not to control it.
  Interventions: Other: Self-treatment by way of Occipivot®

INTERVENTIONS:
Other: Manual technique of sub-occipital inhibition
  Arms: Manual technique of sub-occipital inhibition
Other: Self-treatment by way of Occipivot®
  Arms: Self-treatment by way of Occipivot®

SUMMARY:
The cervical spine should work as a functional unit. If hypomobility should exist in any of the segments it would limit the mobility of the spine as a whole. Although it is frequent that certain cervical segments present hypomobility, they are not always related to symptomatology. The effects of inhibition sub-occipital techniques on cervical mobility have not been evaluated.

The objetive of this trials is to assess and compare the effects on cervical mobility, of the manual technique of sub-occipital inhibition by applying pressure and self-treatment by way of Occipivot® cushion, in subjects with no cervical symptomatology but with limited mobility assessed by the flexion-rotation test.

ELIGIBILITY:
Inclusion Criteria:

* Flexion rotation test with less than 32º or asymmetry of 10º between right and left, whenever one of the sides does not exceed physiological C1-C2 ROM (45º)
* Sing the informed consent form.

Exclusion Criteria:

* Inability to tolerate FRT
* Contraindication to manual therapy.
* Cervical treatment during the study.
* Poor language and communication skills making difficult to undertand the informed consent.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline in Range of movement in Upper Cervical Spine | 15 minutes after intervention
  Flexion-rotation test measured by CROM device

SECONDARY OUTCOMES:
Change in baseline in Range of motion of cervical spine | 15 minutes after intervention
Change in baseline in Upper cervical spine range of motion | 15 minutes after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investgación en Fisioterapia. Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No